CLINICAL TRIAL: NCT01944566
Title: Microbial Community Transplantation on the Armpit in Order to Reduce the Malodour Generation on Armpit.
Brief Title: Microbial Community Transplantation on the Armpit.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013/681
Record Dates: First submitted 2013-09-12; First posted 2013-09-17 (Estimated); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Heavy, Bad Odour From Armpit

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- heavy armpit odour (Experimental): subjects with heavy armpit odour
  Interventions: Biological: Microbial transplant

INTERVENTIONS:
Biological: Microbial transplant — Every subject has 2 armpits; 1 armpit is treated, the other one is not treated. There is a microbial transplant from armpit bacteria.

SUMMARY:
The malodour generation of a person's armpit is caused by the bacteria thriving on that armpit. In order to alter or reduce once bad body odour, the living microbial community on the armpit of a non-malodorous person will be transmitted (or up scaled and transmitted) to the armpit of a malodorous person. The odour is evaluated by a trained smelling panel, the bacteria living on the armpit is examined by means of molecular techniques. The microbial transplantation and its follow-up happens under the supervision of a medical doctor.

ELIGIBILITY:
Inclusion Criteria:

* bad armpit odour

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Reduction of bad odour of the armpit. | 24 evaluations in approximately 10 weeks.
  Odour evaluation by a trained smelling panel. The measurements take place before (once), during the treatment week (5 times) and after the treatment (2x per week during 2 months).
Molecular characterisation of the bacterial community after microbial transplantation. | 24 evaluations in approximately 10 weeks.
  Microbial evaluation by means of DNA extraction and Denaturing Gradient Gel Electrophoresis. The measurements take place before (once), during the treatment week (5 times) and after the treatment (2x per week during 2 months).

SECONDARY OUTCOMES:
Reduction of bad odour of the armpit over a longer period. | after 4 months
  Odour evaluation by a trained smelling panel.
Reduction of bad odour of the armpit over a longer period. | after 6 months
  Odour evaluation by a trained smelling panel.
Molecular characterisation of the bacterial community after microbial transplantation. | after 4 months
  Microbial evaluation by means of DNA extraction and Denaturing Gradient Gel Electrophoresis.
Molecular characterisation of the bacterial community after microbial transplantation. | After 6 months
  Microbial evaluation by means of DNA extraction and Denaturing Gradient Gel Electrophoresis.

CONTACTS AND LOCATIONS:
Overall Officials: Nico Boon, PhD, Study Chair — University Ghent
Locations (2):
- Belgium (2):
  - Ghent University Hospital, Ghent
  - Ghent University, Ghent